CLINICAL TRIAL: NCT00390065
Title: Follow-Up at 6 Years of a Cohort of Children Born Very Prematurely With Respiratory and Neurodevelopmental Impact of Early Treatment With Inhaled Nitric Oxide
Brief Title: Follow-Up at 6 Years of a Cohort of Children Born Very Prematurely
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maternite Regionale Universitaire (Other)
Responsible Party: Principal Investigator, Jean Michel Hascoet, Professor - Head of Division, Maternite Regionale Universitaire
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MRAP060308
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Premature Birth
Keywords: Follow-up; Premature infants; Nitric Oxide; Respiratory function testing; Neurodevelopmental outcomes
MeSH Terms: conditions — Premature Birth | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: This is a follow-up study, at 6 years of age, of infants randomized in the neonatal period with one other group studied as a reference group (ie 3 groups)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization in the neonatal period. Blinding maintained at the time of the follow-up study
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study group (Experimental): Hypoxemic Respiratory Failure treated by Nitric Oxide;
  Interventions: Drug: Nitric Oxide
- Control (Placebo Comparator): Hypoxemic Respiratory Failure control (Placebo);
  Interventions: Drug: Nitric Oxide
- Reference (No Intervention): Reference (Non hypoxemic respiratory failure)

INTERVENTIONS:
Drug: Nitric Oxide — Early low dose (5ppm) NO inhalation Placebo
  Other Names: Reference group (non hypoxemic infants)
  Arms: Control; Study group

SUMMARY:
Utilization of nitric oxide (NO) therapy has been related to a trend towards short term improvement in very premature infants. A two year follow-up of children treated soon after birth with NO in the neonatal period, suggests that a significant improvement in neurodevelopmental outcome might occur. This study aims to evaluate follow-up at 6 years, in respiratory and neurodevelopmental outcome, of children born very prematurely, some of them having been treated with nitric oxide in the neonatal period.

DETAILED DESCRIPTION:
Utilization of nitric oxide therapy in the neonatal period has been related to a trend towards short term improvements in respiratory and neurological outcome at 28 days postnatal age or 36 weeks postconceptional age. A two year follow-up in children treated soon after birth with NO in the neonatal period, suggests that a significant improvement in neurodevelopmental outcome might occur. No long term evaluation on respiratory outcome has yet been done. This study aims to evaluate respiratory and neurodevelopmental outcome at 6 years of age in children born very prematurely, some of them having had Nitric Oxide as a rescue treatment for respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All infants included at birth in a randomized controlled trial using early nitric oxide therapy

Exclusion Criteria:

* Parental refusal

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function testing | at 7 years postnatal age

SECONDARY OUTCOMES:
Neurodevelopmental and Cognitive outcomes | at 7 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, MD, Study Director — University of NANCY, France; Isabelle RM HAMON, MD, PhD, Principal Investigator — Maternite Regionale Universitaire
Locations (2):
- France (2):
  - Maternite Regionale Universitaire, Nancy
  - CHU Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Hascoet JM, Fresson J, Claris O, Hamon I, Lombet J, Liska A, Cantagrel S, Al Hosri J, Thiriez G, Valdes V, Vittu G, Egreteau L, Henrot A, Buchweiller MC, Onody P. The safety and efficacy of nitric oxide therapy in premature infants. J Pediatr. 2005 Mar;146(3):318-23. doi: 10.1016/j.jpeds.2004.10.019. PMID 15756211
- [Background] Deforge H, Andre M, Hascoet JM, Toniolo AM, Demange V, Fresson J. [Cognitive development and attention performances at school age of "normal" prematurely born children]. Arch Pediatr. 2006 Sep;13(9):1195-201. doi: 10.1016/j.arcped.2006.05.015. Epub 2006 Jul 7. French. PMID 16824742
- [Derived] Hamon I, Varechova S, Vieux R, Ioan I, Bonabel C, Schweitzer C, Hascoet JM, Marchal F. Exercise-induced bronchoconstriction in school-age children born extremely preterm. Pediatr Res. 2013 Apr;73(4 Pt 1):464-8. doi: 10.1038/pr.2012.202. Epub 2012 Dec 26. PMID 23269119